CLINICAL TRIAL: NCT02487043
Title: A Telephone-based Case-management Intervention for Caries Prevention in Children With Severe Early Childhood Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Eastmaninstitutet (Other)
Responsible Party: Principal Investigator, Göran Dahllöf, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr 1-314/2013 SOF, KI
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Early Childhood Caries
Keywords: Caries prevention; Early Childhood Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dental health coaches (Experimental): Telephone-based case-management intervention. Contact with families every 2 weeks during one year. Including motivational interviewing, support for dental preventive measures at home, answer questions, care coordination) + conventional protocol (Fluoride prevention program)
  Interventions: Behavioral: A telephone-based case-management intervention
- Control group (No Intervention): Conventional protocol (Fluoride prevention program) and follow-up as usual

INTERVENTIONS:
Behavioral: A telephone-based case-management intervention — Regular Telephone support delivered by Health coaches
  Arms: Dental health coaches

SUMMARY:
Despite improvements in oral health among children, children living in areas characterized by low socio-economic status still have a significant disease burden with regard to dental caries. Special efforts to prevent disease development in this group of children have been unsuccessful. Small children with extensive treatment needs often have limited abilities to cooperate and to provide quality dental care in this patient group, general aneaethesia (GA) may often be the treatment modality of choice. Preschool children treated under general anesthesia have significantly higher caries prevalence (deft and defs), apical parodontitis and infection due to pulpal necrosis. They also have significantly more emergency visits and previous use of treatment under sedation.

This study aim to test the hypothesis, that a telephone based case management intervention for children with severe early childhood caries can prevent further caries development in preschool children who are treated under general anesthesia for severe early childhood caries.

DETAILED DESCRIPTION:
Consecutive children (n=130) who are referred to the departments of pediatric dentistry at Eastman Dental Institute, Public Dental Service and Dental Medicine, Karolinska Institutet, who fulfill inclusion criteria are invited to participate in the study. This is done during the visits preceding the anesthetic evaluation of the patient. Parents will be given written information about the study. During the last visit preceding the GA, a contact is established between dental health coach and family. During this visit the aim of the project is explained and an agreement is signed and informed consent is obtained from the parents only (the parents are the target for this intervention, it is they who perform the preventive oral health measures and supports the child). During this interview, the parents will also answer a structured interview measuring level of self-efficacy and well as their thoughts on dental health care as well as why the situation has occurred. After the initial interview patients are assigned to either intervention group (dental health coach group) or to a control group.

The dental healthcoach will keep in close contact with the intervention group, and by telephone based support provide information, support parental self-efficacy, motivate the family to keep preventive measures that have been individually agreed on, motivate parents to keep preventive appointments and to provide tools for caries prevention.

A follow-up visit is scheduled after 1 year. Parents who decline participation in the program will receive treatment as usual and will be followed for 1 year.

Patients in the control group will receive treatment as usual. This means recall visits to the dental clinic within 3 months after the procedure, reinforcing the individually tailored preventive program. Recall visits after that are scheduled based on treatment needs. A follow-up visit is scheduled after 1 year.

Caries will be diagnosed at baseline ( during GA) and progression will be monitored according to ICDAS after 12 and 24 months. Plaque and gingivitis will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Pre-school children < 6 years of age
* Severe childhood caries
* treated under general anesthesia in Stockholm County Council during a one year period.

Exclusion Criteria:

* Medically compromised children
* Children with learning disabilities

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in New carious lesion (decayed surfaces and decayed teeth) at 12 and 24 months | 12 months, 24 months
  decayed surfaces (dmfs) and decayed teeth (dmft)

SECONDARY OUTCOMES:
Dental attendance | 12 months
  number of visits to dental health care during the observation period, number of unscheduled appointments, number of missed and cancelled appointments
oral health related quality of life | 12 months
  Validated scale OHRQoL, subscales FIS and P-CPQ will be used
Dental Anxiety among parents | 12 months
  Dental Anxiety Scale, DAS
Parental Stress | 12 months
  The Swedish Parenthood Stress Questionnaire - SPSQ
Dental beliefs among parents | 12 months
  Swedish version of the revised Dental Beliefs Survey (DBS-R)

OTHER OUTCOMES:
Dental health coaches' experiences of their role | 18 months
  Questioners and focus groups will be used to understand the experience of the health coach in order to refine the intervention in future projects

CONTACTS AND LOCATIONS:
Overall Officials: Göran Dahllöf, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No
Data collected only for this study

REFERENCES:
- [Derived] Brannemo I, Levinsson A, Hasselblad T, Dahllof G, Tsilingaridis G. Parental psychosocial factors and children's oral health-related quality of life: Data from a caries prevention study with phone-based support. BMC Oral Health. 2025 Jan 18;25(1):94. doi: 10.1186/s12903-025-05446-z. PMID 39827351